CLINICAL TRIAL: NCT00676806
Title: A Phase II Study of Umbilical Cord Blood Transplantation Following Myeloablative or Reduced-Intensity Conditioning
Brief Title: A Phase II Study of Umbilical Cord Blood Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCBT001
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Aplastic Anemia
Keywords: Umbilical cord blood transplantation; full ablation conditioning; reduced intensity conditioning
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Anemia, Aplastic | interventions — Cyclophosphamide; fludarabine phosphate; Busulfan; Ficusin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myeloablative conditioning (Experimental): Umbilical cord blood for hematopoietic rescue following myeloablative conditioning
  Interventions: Biological: Umbilical Cord Blood After Myeloablative Conditioning
- Reduced intensity conditioning (Experimental): Umbilical cord blood for hematopoietic rescue following non-myeloablative conditioning
  Interventions: Biological: Umbilical Cord Blood After Reduced-Intensity Conditioning

INTERVENTIONS:
Biological: Umbilical Cord Blood After Myeloablative Conditioning — cyclophosphamide (60mg/m2 days -6 & -5), fludarabine (25 mg/m2 days -7, -6, & -5) and total body irradiation (days -3, -2, & -1, total 1200 cGy) followed by cord blood infusion on day 0.
  Other Names: Cytoxan; TBI; Fludara; Busulfex; UCBT
  Arms: Myeloablative conditioning
Biological: Umbilical Cord Blood After Reduced-Intensity Conditioning — Extracorporeal Photopheresis (days -8 & -7), cyclophosphamide 50 mg/kg (day -6) pentostatin 4 mg/kg/d (continuous infusion days -5 & -4), total body irradiation (days -3 & -2, total 600cGy) followed by Umbilical Cord Blood Infusion day 0.
  Other Names: Psoralen; Cytoxan; Nypent; TBI; UCBT
  Arms: Reduced intensity conditioning

SUMMARY:
This study is designed to determine whether Umbilical Cord Transplantation (UCB) can be substituted for adult bone marrow cells in the standard stem cell transplant regimens used at this hospital for subjects who do not have stem cell donors.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (SCT) following myeloablative and non-myeloablative conditioning therapy has proven curative treatment for a number of inherited and acquired hematologic disorders. The success of allogeneic transplantation is largely determined by compatibility between donor and recipient, which predicts the risk of fatal graft-versus-host disease (GVHD). Unfortunately, less than one third of patients needing an allogeneic transplant have an available compatible donor in their family. Registries have been established to match patients with compatible volunteer (unrelated) donors, but many patients, and in particular minority patients, still lack stem cell donors.

Umbilical cord blood (UCB) is a rich source of hematopoietic stem cells, which is readily available from the placenta following childbirth. Blood banks have been established in the United States and abroad to collect, process and store UCB for use in allogeneic transplantation. To date, more than 2000 UCB transplants have been performed in adults and children around the world.

Rationale for use of Umbilical Cord Blood in Transplantation

UCB has a number of proven and theoretical advantages as an alternative source of hematopoietic stem cells for transplantation:

1. Placental or umbilical cord blood is an abundantly available source of stem cells, which is currently discarded and can be harvested at no risk to the mother or infant.
2. Important infectious agents, particularly CMV, are much less common in the newborn than adults, and are less likely to contaminate UCB collections.
3. UCB collections, typed, cryopreserved and banked, are available on demand, eliminating delays and uncertainties that now complicate marrow collection from unrelated donors. At present, UCB can be delivered for infusion within days of the initiation of a search. This compares with a median of 3 months from search to delivery of stem cells through the registries of volunteer adult donors.
4. The intensity of graft-versus-host reactivity of fetal lymphocytes appears to be less than that of adult cells and consequently fetal lymphocytes are more tolerant of HLA incompatibility. Published studies have shown that transplantation of UCB matched at 4-5/6 antigens results in a comparable incidence of GVHD to transplantation of unrelated stem cells fully matched at 6/6 antigens.
5. Frozen UCB can be easily shipped, stored at the treating institution, and thawed for use when needed, compared to freshly donated stem cells which have a limited shelf-life of one day or less, necessitating coordination between harvesting surgeons, transportation, and transplantation teams.

This research study has been designed for people who have been diagnosed with a blood tumor, which has not responded to treatment or has recurred, a bone marrow failure state such as aplastic anemia, or one of certain inherited metabolic disorders; and whose doctor feels the best treatment is an allogeneic stem cell transplant (alloSCT) but a related or unrelated adult donor is not available. Instead, a single unit of umbilical cord blood (UCB) will be used as the source of the subject's immune system. This study is designed to determine whether a single unit of UCB can be substituted for adult bone marrow cells in the standard stem cell transplant regimens used at this hospital for subjects who do not have stem cell donors.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting eligibility criteria for unrelated allogeneic stem cell transplantation may be considered for participation on this clinical trial if and only if they meet each of the following criteria:

* Patients must have one of the following diagnoses
* Relapsed or refractory hematologic malignancy, or
* High risk hematologic malignancy in first remission, or
* Refractory acquired marrow failure state, or
* Inherited disorder of metabolism or marrow failure state without alternative curative therapy.
* Patients must not have a 6/6 or 5/6 HLA-matched related donor.
* Patients must not have a HLA-A, -B and -DRB1 high resolution matched unrelated donor following registry search, or cannot (in the opinion of the treating physician) wait the median 3 months to receive a MUD unit.
* Patients must demonstrate an ability to understand and willingness to sign the informed consent document

Patients considered for myeloablative conditioning must satisfy the following additional criteria:

* Patients must be up to age 55 (inclusive)
* Patients must have serum direct bilirubin ≤ 2.0 mg/dl and transaminases ≤ 2x institution upper limit of normal
* Patients must have serum creatinine ≤ 2 mg/dl with creatinine clearance ≥ 60 ml/min (either calculated or measured).
* Patients must have MUGA scan or echocardiogram normal for the institution, but not less than 45% left ventricular ejection fraction and no clinical evidence of cardiac dysfunction.
* Patients must have an ECOG performance status of 0 or 1 (see Appendix C).
* Patients must have adequate pulmonary function when corrected for hemoglobin and alveolar volume as evidenced by a diffusion capacity and FEV1 > 50% of predicted.

Patients considered for reduced-intensity conditioning must satisfy the following additional criteria:

* Patients must not be candidates for myeloablative conditioning due to any one of the following: Prior myeloablative stem cell transplantation, Age > 50, Co morbid illness
* In opinion of treating physician, unable to comply with or withstand rigors of myeloablative conditioning
* Patients with leukemia must have circulating and bone marrow blast counts < 5%, all other patients must have chemotherapy responsive disease
* Patients must be between the ages of 18 and 70 (inclusive)
* Patients must have serum direct bilirubin ≤ 2.0 mg/dL and transaminases ≤ 3x institution upper limit of normal
* Patients must have creatinine clearance ≥ 30 ml/min (either calculated or measured).
* Patients must have MUGA scan or echocardiogram documenting left ventricular ejection fraction of no less than 35% and no clinical evidence of cardiac dysfunction.

Patients must have an ECOG performance status of 0 or 1 (see Appendix C).

Patients must have adequate pulmonary function when corrected for hemoglobin and alveolar volume as evidenced by a diffusion capacity and FEV1 ≥ 40% of predicted.

Exclusion Criteria:

Patients are ineligible for participation on this trial if they meet any of the following criteria:

* Patients with a history of myocardial infarction within the preceding 6 months, significant arrhythmia within the preceding 3 months, uncontrolled hypertension or congestive heart failure are ineligible.
* Patients with unstable angina are not eligible.
* Pregnant or lactating women are ineligible.
* Male and female patients who do not agree to practice approved methods of birth control for the duration of the study are ineligible.
* Patients with uncontrolled infection are ineligible.
* Patients who are HIV positive or have evidence of chronic viral hepatitis are ineligible.
* Patients unable to comply with requirements for compliance with therapeutic plan and/or scheduled evaluations

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-07; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Klein, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject signed consent but did not receive a transplant, so was dropped from the study and was not assigned to either arm.
Groups:
- Myeloablative Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following myeloablative conditioning
  Umbilical Cord Blood Transplantation After Myeloablative Conditioning: Fully-myeloablative Conditioning Regimen: cyclophosphamide (60mg/m2 days -6 & -5), fludarabine (25 mg/m2 days -7, -6, & -5) and total body irradiation (days -3, -2, & -1, total 1200 cGy) followed by cord blood infusion on day 0.
- Reduced Intensity Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following non-myeloablative conditioning
  Umbilical Cord Blood Transplantation After Reduced-Intensity Conditioning: Reduced Intensity Conditioning Regimen: Extracorporeal Photopheresis (days -8 & -7), cyclophosphamide 50 mg/kg (day -6) pentostatin 4 mg/kg/d (continuous infusion days -5 & -4), total body irradiation (days -3 & -2, total 600cGy) followed by Umbilical Cord Blood Infusion day 0.
Period: Overall Study
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (8.1) | 62.6 (2.3) | 52.8 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neutrophil Engraftment
Description: Number of participants with neutrophil engraftment receiving umbilical cord blood for hematopoietic rescue following myeloablative or non-myeloablative conditioning
Time Frame: +45 and 90 days
Population: Only 2 subjects were evaluable from each group at the +45 day mark. The same number were evaluable at the +90 day mark.
Measure: Number; unit: participants
Groups:
- Myeloablative Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following myeloablative conditioning.
  2/2 evaluable subjects engrafted at +45 and +90 days.
- Reduced Intensity Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following non-myeloablative conditioning
  1/2 evaluable subjects engrafted at +45 and +90 days.
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Number analyzed (Participants) | 2 | 2
participants | 2 | 1

2. Secondary Outcome: Proportion of Subjects With Platelet Engraftment
Description: Proportion of patients engrafting by days +45, +90, and +180.
Time Frame: +45, 90, and 180 days
Measure: Number; unit: participants
Groups:
- Myeloablative Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following myeloablative conditioning.
- Reduced Intensity Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following non-myeloablative conditioning
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Number analyzed (Participants) | 2 | 2
participants
  Platelet Engraftment +45 days | 0 | 2
  Platelet Engraftment +90 days | 0 | 0
  Platelet Engraftment +180 days | 1 | 0

3. Secondary Outcome: Incidence of Acute GVHD
Time Frame: Day +100
Measure: Number; unit: participants
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Number analyzed (Participants) | 3 | 3
participants | 1 | 0

4. Secondary Outcome: Infectious Complications in UCB Recipients.
Time Frame: Day +100
Measure: Number; unit: participants
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Number analyzed (Participants) | 3 | 3
participants | 3 | 3

5. Secondary Outcome: Incidence of Chronic GVHD
Time Frame: After Day +100
Population: No subject receiving reduced intensity conditioning was evaluable for the event of chronic GVHD (0/3 subjects survived to day +100)
Measure: Number; unit: participants
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Number analyzed (Participants) | 2 | 0
participants | 1 |

6. Secondary Outcome: Compare Rates of Complications Between Patients Receiving Ablative vs. Non-myeloablative Conditioning Prior to UCB Transplantation
Description: Composite endpoint of GVH or infection. Too few events to compare between arms.
Time Frame: +180 days
Measure: Number; unit: events
Groups:
- Myeloablative Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following myeloablative conditioning.
  2/2 evaluable subjects engrafted at +45 and +90 days. 3 evaluable subjects for toxicity.
- Reduced Intensity Conditioning: Patients receiving umbilical cord blood for hematopoietic rescue following non-myeloablative conditioning
  1/2 evaluable subjects engrafted at +45 and +90 days. 3 evaluable subjects for toxicity.
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Number analyzed (Participants) | 3 | 3
events | 5 | 3

ADVERSE EVENTS:
Arm/Group | Myeloablative Conditioning | Reduced Intensity Conditioning
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Conditioning (N=3) | Reduced Intensity Conditioning (N=3)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Gastrointestinal GVHD (Immune system disorders) | 2 (2) | 0 (0)
Thrombotic microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Conditioning (N=3) | Reduced Intensity Conditioning (N=3)
Skin Nodules (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) — Likely d/t severe medical illness, renal failure, and medication

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes